CLINICAL TRIAL: NCT01832038
Title: A Multi-center, Open-label, Uncontrolled, Long-term, Extension Study to Evaluate the Safety and Efficacy of Lacosamide as Adjunctive Therapy in Japanese and Chinese Adults With Partial-onset Seizures With or Without Secondary Generalization
Brief Title: Study to Evaluate the Safety, Tolerability, and Efficacy of Long-term Adjunctive Therapy With Lacosamide in Adults With Partial-onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Collaborators: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0009
Record Dates: First submitted 2013-03-28; First posted 2013-04-15 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Epilepsy; Partial-onset Seizures
Keywords: Lacosamide; Epilepsy; Partial-onset Seizures
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (Experimental): Lacosamide treatment of 100 - 400 mg/day for long-term
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Strength: Lacosamide (LCM) 50 mg, LCM 100 mg
  Formulation: Tablet
  Frequency: twice daily during the study period (until the date of approval)
  At the completion of EP0008 [NCT01710657], all subjects who choose to enroll in EP0009 will be taking a dose of Lacosamide 200 mg/day. At the beginning of EP0009, the investigator may maintain the LCM dose or increase or decrease the dose. During the Treatment Period, the investigator will be allowed to increase or decrease the dose of LCM to optimize tolerability and seizure reduction. The LCM dose may be decreased to 100 mg/day or increased, no faster than 100 mg/day per week, up to 400 mg/day.
  Other Names: Vimpat

SUMMARY:
The purpose of this trial is to evaluate the safety and tolerability of long-term administration of Lacosamide at doses up to 400 mg/day in Japanese and Chinese adults with Epilepsy who have completed the Treatment and Transition Period of EP0008 [NCT01710657]

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed the Treatment and Transition Period of EP0008 [NCT01710657]

Exclusion Criteria:

* Subjects who withdrew from EP0008 [NCT01710657]

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2013-03-26 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (67):
- China (30):
  - 86026, Beijing
  - 86027, Beijing
  - 86015, Changchun
  - 86005, Chengdu
  - 86032, Chengdu
  - 86006, Chongqing
  - 86031, Dalian
  - 86007, Guangzhou
  - 86008, Guangzhou
  - 86009, Guangzhou
  - 86013, Guangzhou
  - 86016, Guangzhou
  - 86014, Hangzhou
  - 86010, Harbin
  - 86019, Jinan
  - 86004, Kunming
  - 86011, Nanchang
  - 86012, Nanchang
  - 86028, Nanjing
  - 86003, Qingdao
  - 86001, Shanghai
  - 86023, Shanghai
  - 86025, Shanghai
  - 86020, Shijiazhuang
  - 86022, Suzhou
  - 86002, Taiyuan
  - 86018, Wuhan
  - 86024, Wuhan
  - 86017, Xi'an
  - 86029, Xiamen
- Japan (37):
  - 81056, Asaka
  - 81013, Fukuoka
  - 81054, Fukuoka
  - 81057, Hachinohe
  - 81027, Hamamatsu
  - 81004, Himeji
  - 81018, Hiroshima
  - 81019, Iwanuma
  - 81012, Kagoshima
  - 81033, Kitakyushu
  - 81017, Kobe
  - 81024, Kodaira
  - 81010, Kokubunji
  - 81032, Kōshi
  - 81014, Kurume
  - 81047, Kyoto
  - 81035, Nagakute
  - 81028, Nagoya
  - 81029, Nagoya
  - 81040, Nara
  - 81007, Neyagawa
  - 81002, Niigata
  - 81005, Okayama
  - 81011, Saitama
  - 81042, Sakai
  - 81025, Sapporo
  - 81053, Sapporo
  - 81009, Sayama
  - 81021, Shimotsuke
  - 81022, Shimotsuke
  - 81026, Shinjuku
  - 81003, Shizuoka
  - 81023, Suita
  - 81051, Suita
  - 81006, Toyonaka
  - 81050, Ube
  - 81001, Yamagata

REFERENCES:
- [Result] Inoue Y, Liao W, Wang X, Du X, Tennigkeit F, Sasamoto H, Osakabe T, Hoshii N, Yuen N, Hong Z. Safety and efficacy of adjunctive lacosamide in Chinese and Japanese adults with epilepsy and focal seizures: A long-term, open-label extension of a randomized, controlled trial. Epilepsy Res. 2021 Oct;176:106705. doi: 10.1016/j.eplepsyres.2021.106705. Epub 2021 Jun 29. PMID 34246118
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in March 2013 and concluded in July 2019.
Pre-assignment Details: Participant Flow refers to the Safety Set.
Groups:
- Lacosamide: At the completion of EP0008 [NCT01710657], all participants who enrolled in EP0009 were administered a dose of 200 mg/day lacosamide (LCM). The LCM dose may have been decreased to 100 mg/day or increased, no faster than 100 mg/day per week, up to 400 mg/day, at the investigator's discretion.
Period: Overall Study
Arm/Group | Lacosamide
Started | 473
Completed | 238
Not Completed | 235
Not completed — Death | 5
Not completed — Adverse Event | 50
Not completed — Lack of Efficacy | 81
Not completed — Protocol Violation | 7
Not completed — Lost to Follow-up | 10
Not completed — Withdrawal by Subject | 49
Not completed — Visit non-compliance | 2
Not completed — Subject refused to return visit | 2
Not completed — Not convenient to come back to site | 2
Not completed — Participant was asked to quit | 5
Not completed — Back home | 1
Not completed — Pregnancy | 1
Not completed — Low compliance | 3
Not completed — Prohibit procedure | 2
Not completed — Not possible to visit the hospital | 1
Not completed — Changes of implementation system | 3
Not completed — Plan to pregnancy | 7
Not completed — Bad mood and has suicidal thought | 1
Not completed — Prohibited concomitant medication | 1
Not completed — Pregnancy and abortion in EP0008 study | 1
Not completed — Subject considered the efficacy was poor | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set (SS) which consisted of all enrolled participants in EP0009 who took at least 1 dose of lacosamide (LCM) in EP0009.
Arm/Group | Lacosamide
Number analyzed (Participants) | 473
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39
  Between 18 and 65 years | 432
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (12.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 259
  Female | 214
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 350
  Japanese | 123

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Adverse Event Reported Spontaneously by the Subject or Observed by the Investigator From Baseline Until the End of Study Visit
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From Visit 1 (Week 0) up to approximately Week 323
Population: The Safety Set (SS) included all enrolled participants in EP0009 who took at least 1 dose of LCM in EP0009.
Measure: Count of Participants; unit: Participants
Groups:
- Lacosamide (SS): At the completion of EP0008 [NCT01710657], all participants who enrolled in EP0009 were administered a dose of 200 mg/day LCM. The LCM dose may have been decreased to 100 mg/day or increased, no faster than 100 mg/day per week, up to 400 mg/day, at the investigator's discretion. Participants formed the Safety Set (SS).
Arm/Group | Lacosamide (SS)
Number analyzed (Participants) | 473
Participants | 410

2. Primary Outcome: Number of Participants That Withdrew Due to Adverse Events From Baseline Until the End of Study Visit
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment and led to the withdrawal of the participants from the study. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From Visit 1 (Week 0) up to approximately Week 323
Population: The Safety Set (SS) included all enrolled participants in EP0009 who took at least 1 dose of LCM in EP0009.
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide (SS)
Number analyzed (Participants) | 473
Participants | 51

3. Secondary Outcome: Percent Change in Partial-onset Seizure Frequency Per 28 Days From Baseline of Study EP0008 [NCT01710657] Until the End of Study Visit in Study EP0009
Description: The percent change from Baseline to the Treatment Period was calculated as {[(Seizure frequency per 28 days during the Treatment Period) minus (Seizure frequency per 28 days during Baseline Period)] divided by (Seizure frequency per 28 days during Baseline Period)} multiplied by 100. Baseline was defined as the Baseline Period of study EP0008 [NCT01710657].
Time Frame: From Visit 1 in study EP0008 [NCT01710657] up to approximately Week 323 in study EP0009
Population: The Full Analysis Set (FAS) included all study participants from the SS who had at least 1 day with available seizure diary data in study EP0009.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Lacosamide (FAS): At the completion of EP0008 [NCT01710657], all participants who enrolled in EP0009 were administered a dose of 200 mg/day LCM. The LCM dose may have been decreased to 100 mg/day or increased, no faster than 100 mg/day per week, up to 400 mg/day, at the investigator's discretion. Participants formed the Full Analysis Set (FAS).
Arm/Group | Lacosamide (FAS)
Number analyzed (Participants) | 471
Percent change | -44.47 (55.82)

4. Secondary Outcome: Percentage of Participants With 50 % Response Rate in Partial-onset Seizure Frequency Per 28 Days From Baseline of Study EP0008 [NCT01710657] Until the End of Study Visit in Study EP0009
Description: A responder is a subject experiencing a greater than or equal to (≥) 50 % reduction in partial-onset seizure frequency per 28 days from baseline. Baseline was defined as the Baseline Period of study EP0008 [NCT01710657].
Time Frame: From Visit 1 in study EP0008 [NCT01710657] up to approximately Week 323 in study EP0009
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide (FAS)
Number analyzed (Participants) | 471
percentage of participants | 57.1

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Visit 1 (Week 0) up to approximately Week 323
Arm/Group | Lacosamide (SS)
All-Cause Mortality (participants affected / at risk) | 6/473
Serious Adverse Events (participants affected / at risk) | 83/473
Other Adverse Events (participants affected / at risk) | 343/473
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (SS) (N=473)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Hamartoma (Congenital, familial and genetic disorders) | 1 (1)
Blindness unilateral (Eye disorders) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastritis atrophic (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Hypertrophic anal papilla (Gastrointestinal disorders) | 1 (1)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Bacterial prostatitis (Infections and infestations) | 1 (1)
Chronic sinusitis (Infections and infestations) | 2 (2)
Encephalitis viral (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Orchitis (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Retroperitoneal infection (Infections and infestations) | 1 (1)
Tuberculosis of genitourinary system (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 2 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (3)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 1 (3)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 2 (2)
Jaw fracture (Injury, poisoning and procedural complications) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Meigs' syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian germ cell teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2)
Complex partial seizures (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 3 (3)
Epilepsy (Nervous system disorders) | 10 (10)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1)
Intracranial haematoma (Nervous system disorders) | 1 (1)
Partial seizures with secondary generalisation (Nervous system disorders) | 1 (1)
Seizure cluster (Nervous system disorders) | 1 (2)
Status epilepticus (Nervous system disorders) | 11 (13)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2)
Temporal lobe epilepsy (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Visual field defect (Nervous system disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Epileptic psychosis (Psychiatric disorders) | 3 (3)
Hallucination (Psychiatric disorders) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abortion induced (Surgical and medical procedures) | 3 (3)
Wisdom teeth removal (Surgical and medical procedures) | 2 (2)
Varicose vein (Vascular disorders) | 1 (1)
Venous occlusion (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (SS) (N=473)
Vision blurred (Eye disorders) | 22 (29)
Abdominal pain upper (Gastrointestinal disorders) | 28 (57)
Diarrhoea (Gastrointestinal disorders) | 41 (64)
Nausea (Gastrointestinal disorders) | 30 (46)
Toothache (Gastrointestinal disorders) | 38 (47)
Vomiting (Gastrointestinal disorders) | 37 (66)
Pyrexia (General disorders) | 41 (53)
Gastroenteritis (Infections and infestations) | 27 (36)
Nasopharyngitis (Infections and infestations) | 156 (510)
Pharyngitis (Infections and infestations) | 22 (38)
Upper respiratory tract infection (Infections and infestations) | 99 (208)
Contusion (Injury, poisoning and procedural complications) | 27 (37)
Dizziness (Nervous system disorders) | 125 (318)
Headache (Nervous system disorders) | 77 (177)
Somnolence (Nervous system disorders) | 41 (80)
Insomnia (Psychiatric disorders) | 26 (32)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (43)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 27 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2013-03-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT01832038/Prot_000.pdf
  • Statistical Analysis Plan (2014-09-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT01832038/SAP_001.pdf